CLINICAL TRIAL: NCT05597917
Title: Phase III Study Comparing Trabectedin (T) Versus T Plus tTF-NGR to Entrap T Inside the Tumor in Patients With Metastatic and/or Refractory Soft Tissue Sarcoma (STS)
Brief Title: tTF-NGR Randomized Study - STS
Acronym: TRABTRAP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universität Münster (Other)
Collaborators: Anturec Pharmaceuticals GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WWU19_0007; 2024-516392-33-00 (EU CTIS Number); 2020-005858-21 (EudraCT Number)
Record Dates: First submitted 2021-06-14; First posted 2022-10-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Soft Tissue Sarcoma
Keywords: tTF-NGR; vascular targeting; CD13; aminopeptidase N; Trabectedin
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Standard chemotherapy with trabectidin (in-label) (Active Comparator): Patients will receive standard trabectedin 1.5 mg/m2 as a 24-hour central intravenous (IV) infusion on day 1, q d 22 x until disease progression or contraindications against further application.
  Interventions: Drug: Trabectedin
- Arm 2: tTF-NGR added to standard trabectedin (Experimental): Patients will receive standard trabectedin according to arm 1 plus 0.5 mg/m2 tTF-NGR (1-hour ratecontrolled infusion, port central venous access, 0.9 % NaCl ad 100 mL) on days 2 and 3 following each trabectedin cycle (within 1 hour interval between end of trabectedin infusion and tTF-NGR: e.g.: trabectedin on monday 8 am to tuesday 8 am followed by tTF-NGR on tuesday 9 am and on the following day, q d 22 x until disease progression or contraindications against further application.
  Interventions: Drug: Trabectedin; Biological: tTF-NGR

INTERVENTIONS:
Drug: Trabectedin — Patients will receive standard trabectedin 1.5 mg/m2 as a 24-hour central intravenous (IV) infusion on day 1, q d 22 x until disease progression or contraindications against further application.
  Other Names: Yondelis
Biological: tTF-NGR — Patients will receive standard trabectedin according to arm 1 plus 0.5 mg/m2 of tTF-NGR (1-hour ratecontrolled infusion, port central venous access, 0.9 % NaCl ad 100 mL) on days 2 and 3 following each trabectedin cycle (within 1 hour interval between end of trabectedin infusion and tTF-NGR: e.g.: trabectedin on monday 8 am to tuesday 8 am followed by tTF-NGR on tuesday 9 am and on the following day, q d 22 x until disease progression or contraindications against further application.
  Arms: Arm 2: tTF-NGR added to standard trabectedin

SUMMARY:
In this phase III open label, controlled clinical trial patients with unresectable or metastatic soft-tissue sarcoma after failure of anthracycline-containing first line therapy or with contraindications to these drugs and CD13 positivity in central histology (grade >/= 1+) are treated to evaluate whether tTF-NGR in combination with standard trabectedin chemotherapy prolongs progression-free survival (according to iRECIST), as compared with trabectedin alone. Further objectives are to evaluate the efficacy of tTF-NGR in combination with standard trabectedin chemotherapy with respect to the response rate and overall survival as well as to assess the safety profile of tTF-NGR combined with trabectedin. Before the randomized phase III part of the study, there was a safety run-in part. The final dose of tTF-NGR established as safe in this safety run-in part is 0.5 mg/m2 per day for 2 consecutive days following each trabectedin infusion and is used for the randomized (parallel 1:1; Arm 1: standard trabectedin, Arm 2: standard trabectedin plus tTF-NGR) phase III part of this trail. . Further dose modification for tTF-NGR is possible.

DETAILED DESCRIPTION:
Rationale: tTF-NGR targets CD13 present in tumor-associated vasculature and on tumor cells of the majority of STS tissue samples examined; preclinical data on combination of tTF-NGR with anthracyclines and trabectedin; low competition of targeted or immune therapy in soft tissue sarcoma (STS)

Investigational Medicinal Product: Patients will receive a dose of the Investigational Medicinal Product (IMP) tTF-NGR determined to be safe within the safety run-in cohort of the study as 1-hour rate-controlled infusion (port central venous access, 0.9 % NaCl ad 100 mL) per day for 2 consecutive days following each trabectedin cycle (within 1 hour interval between end of trabectedin infusion and tTF-NGR: e.g.: trabectedin on monday 8 am to tuesday 8 am followed by tTF-NGR on tuesday latest 9 am and on the following day, q d 22 x until disease progression or contraindications against further application.

Indication: Unresectable or metastatic STS after failure of anthracycline-containing first line treatment or with contraindications to these drugs; CD13 positivity in central histology (grade >/= 1+)

Primary objective and endpoints: The primary objective of the trial is to evaluate whether tTF-NGR in combination with standard trabectedin chemotherapy given for unresectable or metastatic soft tissue sarcoma after failure of anthracycline-containing first line therapy or with contraindications to these drugs prolongs progression-free survival, as compared with trabectedin alone. The following efficacy endpoint (for the randomized phase III part) will be considered:

- Progression-free survival (PFS) according to iRECIST (Seymour L, Lancet Oncol. 2017) as judged by central radiology in a blinded fashion after end of trial.

Secondary objectives and endpoints: The secondary objective of the trial is to evaluate the efficacy of tTF-NGR in combination with standard trabectedin chemotherapy given for unresectable or metastatic STS after failure of anthracycline-containing first line therapy or with contraindications to these drugs with respect to the response rate and overall survival as well as to assess the safety profile of tTF-NGR combined with trabectedin.

To assess the efficacy, the following measurements will be considered:

* Overall response rate (ORR, consisting of CR and PR)
* Disease control rate (DCR, consisting of CR, PR, and stable disease (SD) for >18 weeks)
* Median progression-free survival (mPFS)
* Median overall survival (mOS)
* Overall survival (OS) rate at 12 and 18 months

To assess the safety profile of tTF-NGR combined with trabectedin (for the phase II and the phase III parts), the following safety endpoints will be considered:

* Adverse Events (AEs) assessment based on CTCAE v.5.0.
* Standard laboratory parameters and pharmacokinetics
* Physical examination findings including assessment of vital signs
* Patient reported outcomes (PRO)

Study design: Open label, randomized, controlled study in subjects with metastatic or refractory soft tissue sarcoma. Approx. 150 patients will be screened, 126 evaluable patients are enrolled and parallel assigned in a 1:1 fashion to one of two different arms, as outlined below. Randomization will be stratified into CD13+ grades 1 and 2 versus CD13+ grade 3 and number of chemotherapy regimen before entry on trial: 1 versus >1.

Safety run-in part:

Before the randomized phase III part of the study, there was a safety cohort of a minimum of 6 patients obtaining at least 2 cycles each of the combination outlined in arm 2 (see below) to confirm safety of this combination (1.5 mg/m2 trabectedin plus a starting dose of 3 mg/m2 tTF-NGR). The patients were treated in-house and in sequence. In case of dose-limiting toxicity (DLT) in one patient of this cohort, a dosemodification protocol for tTF-NGR to 2 mg/m2 was planned, and in case of further tolerability problems in one patient further deescalations in 0.5 mg/m2 steps of tTF-NGR and/or by a reduction of application days were planned. The safety part of the study is completed and the safe dose of tTF-NGR for the randomized phase III part of the study is 0.5 mg/m2 given on days 2 and 3. Since 6 patients tolerated >/= 2 cycles of this dose without DLT, DLT should occur in </= 10 % of the patients treated in arm 2 of the trial. The randomized part of the study is open after approval by the DSMB, Ethics Committee and National Competenent Authority (PEI).

Randaomzied Phase III part:

ARM 1:

Trabectedin 1.5 mg/m2 as a 24-hour central intravenous (IV) infusion on day 1, q d 22 x until disease progression or contraindications against further application.

ARM 2:

Patients will receive standard trabectedin according to arm 1 plus t0.5 mg/m2 tTF-NGR (1-hour ratecontrolled infusion, port central venous access, 0.9 % NaCl ad 100 mL) one days 2 and 3 following each trabectedin cycle (within 1 hour interval between end of trabectedin infusion and tTF-NGR: e.g.: trabectedin on monday 8 am to tuesday 8 am followed by tTF-NGR on tuesday 9 am and on the following day, q d 22 x until disease progression or contraindications against further application. Further dose modification for tTF-NGR is possible (see chapeter 6.1.4 of the protocol).

As the evaluation of the study results is based on an intention-to-treat analysis, all patients after randomization will be part of the efficacy population as evaluated by central iRECIST evaluation after end of study.

Therapy in both arms can be given on an out-patient basis. All patients receive best supportive care (BSC) according to institutional guidelines. Anti-cancer activity (iRECIST modification) will be assessed (clinically and imaging) at week 9 and then every 9 weeks (independent from cycle length or number) until confirmed progression by iRECIST (iCPD). Decision on application of next cycle at week 9 will be clinical. Imaging and clinical based decision will follow. Transfer of pseudonymized imaging pictures (CD, DVD) and imaging results of a patient to the study center has to be performed after each imaging time point.

Safety assessment will be performed on an ongoing basis during study participation, including standard laboratory assessments. The incidence of AEs will be summarized by severity in all patients with at least one study drug intake.

Number of sites, countries and patients: Multicenter, up to 14 active study sites in Germany. 19 patients were treated in the phase II safety part, 126 patients will be randomized in a 1:1 ratio to receive open label Trabectedin (Arm 1) or Trabectedin plus tTF-NGR (Arm 2) in the phase III part.

Target population: Patients (18-75 years) with advanced or metastatic soft-tissue sarcoma after failure of anthracycline-containing first line therapy or with contraindications to these drugs.

ARM 1: Standard chemotherapy with Trabectidin (in-label)

ARM 2: Test product tTF-NGR added to standard Trabectedin

Severity grading: Hematological and chemical laboratory tests, and AEs will be graded based on CTCAE v. 5.0.

Duration of Treatment: Patients will be treated in repeated cycles until definite disease progression (iRECIST; Seymour L, Lancet Oncol. 2017) in the absence of other withdrawal criteria, and as long as neither patient nor investigator requests treatment discontinuation.

Tumor assessments: Detailed tumor assessment visits (clinical and laboratory examinations) after start of therapy are performed before treatment start, at week 9 (+/- 1 week), followed by every 9 weeks (+/- 1 week, independent from cycle length or number) thereafter. Post-study treatment (treatment with another anti-cancer agent) is according to investigator´s choice, but is recorded in the eCRF. At iCPD (confirmed at next tumor assessment after iUPD) tumor assessments will end, but time of death will be recorded for estimation of OS. In case EOT is not determined by iCPD, tumor assessments will go on after EOT until iCPD. Survival status will be collected also for patients withdrawn from the study until death. Transfer of pseudonymized imaging pictures (CD, DVD) and imaging results of a patient to the study center has to be performed after each imaging time point.

Statistical analysis: Safety data of the safety run-in part of the study were evaluated using descriptive statistical methods.

In the primary statistical analysis of the randomized phase III part, the primary endpoint progression-free survival (PFS) according to iRECIST as judged by central blinded radiology will be compared between the two randomized treatment groups (Arm 1 versus Arm 2). The primary statistical analysis will include all randomized patients (full analysis set) and will be performed according to the intention-to-treat principle. A stratified log-rank test with stratification according to the randomization will be applied (two-sided significance level 5%, power 80%) that provides confirmatory statistical evidence.

The timing of the study will be event-driven. The primary statistical analysis will be performed at the time when 106 events in terms of PFS have been observed in total across both treatment groups. This required number of events results from the following sample size calculation. Based on the observed PFS in previous trials, PFS is expected to be exponential, and the expected median PFS is 4.6 months in the control arm (Arm 1) and 8 months in the experimental arm (Arm 2). The corresponding expected hazard ratio is HR=0.575. In a 36 months enrolment period with a rate of 3-4 patients per month, 126 patients will be recruited and randomized. The drop-out process after randomization is expected to be exponential with an up to 25% cumulative drop-out rate at month 24 (competing with the survival process). Follow-up after the last randomized patient is planned to be 12 months, after which it is expected that the required number of 106 events in terms of PFS will have occurred.

The statistical analysis of pre-specified secondary endpoints will be performed with descriptive and inferential statistical methods. Prespecified subgroup analyses will be performed with respect to stratification, L-sarcoma vs. others, FNCLCC grade (2 vs. 3), ECOG performance status (ECOG PS 0 vs. PS 1) and previously obtained Lurbinectedin/Trabectedin versus no such previous exposition. Further exploratory analyses will be performed for other relevant treatment variables (e.g. sex, age, number of treatment cycles).

Safety data will be evaluated and summarized descriptively.

Withdrawal and patient replacement criteria: The patient can withdraw consent for participation in the study at any time without disadvantages for further treatment or prejudice by the therapeutic team. The investigator can withdraw a patient if, in his or her clinical judgment, it is in the best interest of the patient or if the patient cannot comply with the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of all genders (female, male, diverse), with no restriction regarding ethnic or religious background age 18 - 75 years.
2. Patients with advanced or metastatic soft-tissue sarcoma after failure of anthracycline-containing first line therapy (or anthracycline-containing adjuvant therapy within 12 months before entry on study) or with contraindications to these drugs
3. Patients must have histological evidence of high-grade advanced unresectable or metastatic soft tissue sarcoma (grade 2 - 3) according to the FNCLCC grading system. The following tumor types are included:

   * Dedifferentiated liposarcoma
   * Myxoid liposarcoma (high grade)
   * Pleomorphic liposarcoma
   * Adult fibrosarcoma
   * Myxofibrosarcoma (high-grade)
   * Leiomyosarcoma
   * Rhabdomyosarcoma (alveolar, pleomorphic)
   * Angiosarcoma
   * Synovial sarcoma
   * Undifferentiated sarcoma

   Tumor types not listed above may be included upon communication with Coordinating Investigator.

   The following tumor types will not be included:
   * Gastrointestinal stromal tumors (GIST)
   * Epitheloid sarcoma
   * Alveolar soft part sarcoma
   * Desmoplastic small round cell tumor
   * Chondrosarcoma
   * Osteosarcoma
   * Ewing sarcoma (including CIC-rearranged sarcoma and Sarcoma with BCOR alterations)
4. CD13 positivity with a score of ≥ 1 (20) by central pathology (GDI Münster)
5. Patients must have at least one unidimensionally measurable lesion by computed tomography as defined by RECIST criteria 1.1. Other adequate imaging procedures such as MRI are allowed. This lesion should not have been irradiated during previous treatments
6. Life expectancy of at least 3 months
7. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
8. No contraindications for trabectedin (see attachment)
9. Negative serum pregnancy test for females of childbearing potential* within 14 days of starting treatment
10. Informed consent signed and dated to participate in the study
11. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures

    * Women of childbearing potential (WOCBP) must be using, from the screening to 3 months following the last trabectedin (Arm 1) or the last last study drug (Arm 2) administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesteron-only or combined (estrogen- and progesteron-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomized partner or sexual abstinence. Pregnancy test will be repeated monthly. For men contraception methods should be performed for 5 months after the last application of trabectedin (Arm1) or study drug (Arm 2).Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy)

Exclusion Criteria:

1. curative therapy available
2. clinically significant unrelated illness, which in the judgement of the investigators could compromise the patient's ability to tolerate the IMP or be likely to interfere with the study procedures or results
3. immobilized tumor patients (wheel chair etc.) with increased risk for DVT
4. known hypersensitivity reactions to prior application of E. coli-derived material
5. history of coronary heart disease, stroke, transitent ischemic attacks, pulmonary embolism, or deep vein thrombosis. For reason of mechanism of action of tTF-NGR, exclusion of patients with a history of any of the vascular conditions mentioned is important. Clinical suspicion of coronary heart disease must be further checked e.g. by cardiac MRI or myocardial scintigraphy to exclude coronary heart disease.
6. known hereditary syndromes with elevated thromboembolic risk (FV Leiden and prothrombin mutations (G20210A), hereditary antithrombin, protein C and S deficiency, and antiphospholipid syndrome) after one or more clinical thromboembolic events
7. patients with hereditary vascular disorders (such as Klippel-Trenauny-Weber syndrome) with increased thromboembolic risk.
8. patients with a Khorana score of (Khorana AA, et al. J.Clin. Oncol. 2009, 27, 4839-4847, attached to this protocol) of > 3
9. elevated Troponin T hs (> 50 ng/L) or elevated Troponin I hs before entry on study
10. presence of active central nervous system (CNS) disease and/or CNS vascular abnormalities detected by MRI or CT
11. no adequate bone marrow function, absolute neutrophil count (ANC) < 1.0 x 109/L, platelets < 50 x 109/L (for trabectedin actually < 100 x 109/L - to be decided by the investigator on an individual patient basis) and haemoglobin (Hb) < 8.0 g/dl.
12. chronically impaired renal function or creatinine ≥ 2.0 x upper limit of normal (ULN).
13. inadequate liver function (alanine aminotranserase (ALT), aspartate aminotranserase (AST), alkaline phosphatase (ALP) or total bilirubin ≥ 2.5 x ULN) unless due to liver metastasis (decision by the investigator)
14. fibrinogen < 150 mg/dL, and/or International Normalized Ratio (INR) > 1,5 (global coagulation parameters can be discussed with the Coordinating Investigator prior to entry on study)
15. female patients with child-bearing who do not agree to exclusion of potential pregnancy by adequate testing within 48 hours prior to entry on study
16. females of childbearing potential as well as fertile males who do not agree to use a highly effective form of contraception (Pearl Index < 1) during the study and for 3 months (females) following the last trabectedin (Arm 1) or last study drug (Arm 2) administration and 5 months (males) following the last dose of trabectedin (Arm 1) or study drug (Arm 2)
17. women with breast-feeding activity
18. concomitant use of any other investigational agent (agent for which there is currently no approved indication from regulatory authorities) or any other anti-cancer drug
19. concomitant enrolment in another clinical trial interfering with the endpoints of this study.
20. any medical condition which could compromise participation in the study according to the investigator's assessment.
21. prophylactic or therapeutic anticoagulation within the last 3 days
22. presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study
23. concurrent malignancies other than STS, unless the patient has been disease-free for at least 2 years
24. serious, non-healing wound, ulcer or bone fracture; not completed wound healing from previous wounds and/or surgery
25. no central venous port system in place (the option of other central venous access than a port should be discussed with the Coordinating Investigator).

NOTE: Outliers of laboratory values can be disregarded and set aside as exclusion criteria by a Coordinating Investigator´s decision. The conditions for the use of trabectedin as specified in the Summary of Product Characteristics are to be followed according to institutional guidelines for standard of care.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Prolongation of progression-free survival (PFS) according to iRECIST as judged by central radiology in a blinded fashion after end of trial. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The primary objective of the trial is to evaluate whether tTF-NGR in combination with standard trabectedin chemotherapy given for unresectable or metastatic soft tissue sarcoma after failure of anthracycline-containing first line therapy or with contraindications to these drugs prolongs progression-free survival, as compared with trabectedin alone.
  The following efficacy endpoint (for the randomized phase III part) will be considered:
  - Progression-free survival (PFS) according to iRECIST (Seymour L, Lancet Oncol. 2017) as judged by central radiology in a blinded fashion after end of trial.

SECONDARY OUTCOMES:
Evaluation of the efficacy of tTF-NGR in combination with standard trabectedin chemotherapy (OOR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the efficacy, the following measurement will be considered:
  Overall response rate (ORR, consisting of CR and PR)
Evaluation of the efficacy of tTF-NGR in combination with standard trabectedin chemotherapy (DCR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the efficacy, the following measurement will be considered:
  - Disease control rate (DCR, consisting of CR, PR, and stable disease (SD) for >18 weeks)
Evaluation of the efficacy of tTF-NGR in combination with standard trabectedin chemotherapy (mPFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the efficacy, the following measurement will be considered:
  - Median progression-free survival (mPFS)
Evaluation of the efficacy of tTF-NGR in combination with standard trabectedin chemotherapy (mOS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the efficacy, the following measurement will be considered:
  - Median overall survival (mOS)
Evaluation of the efficacy of tTF-NGR in combination with standard trabectedin chemotherapy (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the efficacy, the following measurement will be considered:
  - Overall survival (OS) rate at 12 and 18 months
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (AE) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - Adverse Events (AEs) assessment based on CTCAE v.5.0.
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (Standard laboratory parameters) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - laboratory parameter: Troponin T hs [ng/l]
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (Physical examination: Height) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - Physical examination: Height [m]
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (Physical examination: Weight) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - Physical examination: Weight [kg]
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (Physical examination: Body surface) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - Physical examination: Body surface area [m2]
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (Vital sign: breathing) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - Physical examination: Vital sign: breathing rate by watching and counting [breaths per minute]
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (Vital sign: consciousness) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - Physical examination: Vital sign: consciousness by talking to the patient
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (Vital sign: heart rate) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - Physical examination: Vital sign: heart rate by pulse [beats per minute]
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (Physical examination: ECOG perfomance status) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - Physical examination: ECOG perfomance status
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (ECG) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - ECG (rythm, puls rate, Vector, P Wave, PQ time, QRS Complex, R progression from V1 to V6, QT Interval, PQ time, QRS time, T wave)
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (Echocardiography) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - Echocardiography (diameters of both atria and left and right cardiac chambers at end-diastolic and end-systolic times [mm], ejection fraction [%], wall diameters [mm])
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (PRO) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - Patient reported outcomes (PRO) by EORTC QLQ C30 questionnaire
Evaluation of the safety profile of tTF-NGR combined with standard trabectedin chemotherapy (PK) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To assess the safety profile of tTF-NGR combined with trabectedin the following safety endpoint will be considered:
  - pharmacokinetics: AUC [ng*h/ml]

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schliemann, Prof. Dr., Principal Investigator — University Hospital Muenster (Department of Medicine A), Germany
Locations (9):
- Germany (9):
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - HELIOS Klinikum Berlin-Buch, Berlin
  - TU Dresden Medizinische Fakultät Carl Gustav Carus, Dresden
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsmedizin Mainz, Mainz
  - Klinikum rechts der Isar der technischen Universität München, München
  - LMU Klinikum, Münich
  - University Hospital Muenster, Germany, Münster

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for all primary and secondary outcome measurements will be made available within 6 months of study completion
Supporting Information: Study Protocol
Time Frame: within 6 months of study completion